CLINICAL TRIAL: NCT01826058
Title: Spine Stereotactic Body Radiation Therapy for Metastatic Epidural Spinal Cord: Prospective Phase II Study
Brief Title: Spine Stereotactic Body Radiation Therapy for Metastatic Epidural Spinal Cord Compression
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Samsung Medical Center (Other)
Collaborators: Seoul National University Hospital (Other); Gachon University Gil Medical Center (Other)
Responsible Party: Principal Investigator, Doo Ho Choi, Professor, Department of Radiation Oncology, Samsung Medical Center, Sungkyunkwan University School of Medicine, Samsung Medical Center
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KROG 1316
Record Dates: First submitted 2013-04-03; First posted 2013-04-08 (Estimated); Last update posted 2014-12-02 (Estimated); Status verified 2014-11

CONDITIONS: Spinal Cord Compression
Keywords: Stereotactic body radiation therapy; Radiosurgery
MeSH Terms: conditions — Spinal Cord Compression | interventions — Radiosurgery; Radiation; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Stereotactic body radiation therapy (Experimental): SBRT in one to four fractions
  Irradiated total RT dose to gross tumor volume (GTV) according to fraction size
  * 1 fx: 16 to 24 Gy
  * 2 fx's: 20 to 26 Gy
  * 3 fx's: 21 to 30 Gy
  * 4 fx's: 24 to 36 Gy
  Interventions: Radiation: Stereotactic body radiation therapy

INTERVENTIONS:
Radiation: Stereotactic body radiation therapy
  Other Names: Radiosurgery; SRS; Radiation; Radiotherapy; Metastatic Epidural Spinal Cord Compression; MESCC

SUMMARY:
Metastatic epidural spinal cord compression (MESCC) is a frequent oncologic emergency that requires to be treated promptly. Although direct decompressive surgery is the most effective treatment, surgery is only used in selected patients because most patients have a poor overall condition and short life expectancy. Radiation therapy (RT), therefore, is the most commonly used for patients with MESCC, but conventional RT alone can achieve modest neurologic outcomes.

The hypothesis to use stereotactic body radiation therapy (SBRT) for MESCC is that the rapid decompression of epidural mass, durable local control and subsequently improved neurologic outcomes compared to conventional RT are expected when MESCC is treated with SBRT.

DETAILED DESCRIPTION:
The definition of metastatic epidural spinal cord compression (MESCC)

* MESCC is defined as both an evidence of cord compression by radiologic evaluation and a manifestation of clinical feature at the level of cord compression.
* A cord compression by radiologic evaluation is defined as < 3mm gap between epidural mass and true spinal cord or indentation of thecal sac at the level of clinical feature by MRI.
* Clinical features include any or all of the followings: pain (local or radicular) or motor weakness or sensory change or incontinence.

Simulation -A Computed tomography (CT) scan will be acquired with the use of intravenous contrast and planning MRI will be also performed on the same day of simulation.

Spine SBRT

- One to four sessions of SBRT will be performed.

Follow-up

* Patients need to be assessed at 1 week, 1 month and 3 months after the completion of SBRT and will be followed up at 3 month intervals thereafter.
* Pain score, neurologic examination, adverse events and simple X-ray of involved spine should be evaluated at every follow-up visit.
* MRI of involved spine will be performed at 3 months after the completion of SBRT.

Up to 43 patients will be enrolled in this study in Samsung Medical Center, Seoul National University Hospital, and Gachon University Gil Medical Center.

ELIGIBILITY:
Inclusion Criteria:

* MESCC is present.
* Localized spine metastases (C1 to L5 level); Maximum 3 separate sites and maximum 2 contiguous vertebral bodies
* Performance state before the occurrence of neurologic symptoms : Eastern Cooperative Oncology Group 0-2
* Age ≥20
* MRI within 2 weeks is mandatory
* Paraspinal mass < 5cm in maximum dimension
* Inoperable patients - refused or medically unfit for decompression surgery
* life expectancy > 3 months

Exclusion Criteria:

* Retropulsed bony fragment causing cord compression
* Paraplegia ≥ 48 hours
* Histology preferred to perform the chemotherapy as the first option (e.g. lymphoma, myeloma)

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Estimated)
Dates: Start 2012-10; Primary Completion 2015-06 (Estimated); Study Completion 2015-08 (Estimated)

PRIMARY OUTCOMES:
Neurologic response | 1 month
  * Neurologic response is defined as maintaining grade 4 or more motor power after completing SBRT or as an increase of motor power by at least 1 grade from the baseline motor power.
  * There should no decrease of motor power after completing SBRT.
  * The motor weakness is graded from 0 to 5 by Medical Research Council (MRC) scale.

CONTACTS AND LOCATIONS:
Locations (1):
- Samsung Medical Center, Seoul, South Korea